CLINICAL TRIAL: NCT04197557
Title: The National Survey on Bone Age of Child in China
Brief Title: Bone Age of Chinese Child (BACC)
Acronym: BACC
Status: Completed | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: National Institute for Nutrition and Health Chinese Center for Disease Control and Prevention (Unknown); Beijing pediatric research institute (Unknown)
Responsible Party: Principal Investigator, xiaoguang Cheng, Professor, chairman of Radiology Department, Beijing Jishuitan Hospital
Other Study IDs: JST2019BA
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Bone Development
Keywords: bone age; bone mineral density; X-ray; Chinese child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The bone age of the hand and wrist will be assessed with X-rays in more than 20,000 healthy children age 3-18 years old recruited in 28 sites from 14 province.The bone mineral density (BMD) will be measured as well.

DETAILED DESCRIPTION:
As part of the "National Nutrition and Health Systematic Survey for 0-18 years old Children and Utilization of Survey Findings "(ChiCTR1900022825), more than 20,000 children age 3-18 years old was recruited from 28 sites of 14 provinces within the framework of the ChiCTR190002282 study protocol. The population of this study was proportional to the ChiCTR190002282 study. The X-ray of no-dominant hand and wrist was taken with a mobile X-ray unit with shielding. A step wedge was imaged along the side of the hand at the same time for bone mineral density measurement. The bone age of the hand and wrist was assessed by trained MSK radiologists according to Chinese standard. The bone mineral density of the wrist was measured with radioabsorptiometry (RA). The demographic parameters were collected by the study of ChiCTR190002282 protocol.

ELIGIBILITY:
Inclusion Criteria:

* participants of ChiCTR1900022825 study
* healthy children age 3 to 18 years old.
* willing to participate this study
* Consent by parents

Exclusion Criteria:

* no consent by parents
* under 3 years old

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: As part of the "National Nutrition and Health Systematic Survey for 0-18 years old Children and Utilization of Survey Findings" (ChiCTR1900022825). This population is the subset of the ChiCTR1900022825 study, age 3-18 years old, sample proportion to the general study population. General healthy children age over 3 years old up to 18 years old from the kindergarden, primary school, middle school and high school.
Sampling Method: Probability Sample
Enrollment: 20166 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
the bone age of the wrist and hand | 3 years
  The bone age assessed by radiologist with the hand and wrist X-ray

SECONDARY OUTCOMES:
bone mineral density (BMD) | 3 years
  The bone mineral density (BMD) measured with the wrist and hand X-ray The bone mineral density (BMD) measured with the wrist and hand X-ray calibrated with a step wedge

CONTACTS AND LOCATIONS:
Overall Officials: xiaoguang cheng, MD, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China